CLINICAL TRIAL: NCT00513279
Title: A First Time in Human, Blinded, Randomised, Placebo-Controlled, Two-cohort Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single Oral Escalating Doses of GSK618334 in Healthy Male Volunteers
Brief Title: To Investigate If Single Doses Of GSK618334 Are Safe And To Investigate Blood Levels Of GSK618334
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: DBU107640
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Substance Dependence
Keywords: Safety,; GSK618334; pharmacokinetics,; repeat dose,; tolerability,; pharmacodynamics,; placebo,
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects in Cohort 1 will be randomized to one of the following sequences: ABDFH, BADFH, BDAFH, BDFAH and BDFHA in a 1:1:1:1:1 ratio where A = Placebo, B= GSK618334 dose 1 (2.5 mg), D = GSK618334 dose 3, F = GSK618334 dose 5, H = GSK618334 dose 7. On day 1, subjects will be administered a starting dose of 2.5 milligrams (mg) GSK618334. The planned doses of GSK618334 to be administered in Cohort 1 are 2.5, 25, 100 and 400mg. In each dosing period 2 subjects will receive placebo and 8 subjects will receive GSK618334. Subjects within a cohort will have a washout period of at least two weeks from last dose before receiving another dose.
  Interventions: Drug: GSK618334; Drug: GSK618334 matching placebo tablets
- Cohort 2 (Experimental): Subjects in Cohort 2 will be randomized to one of the following sequences: ACEGI, CAEGI, CEAGI, CEGAI, CEGIA in a 1:1:1:1:1 ratio where A = Placebo, C= GSK618334 dose 2, E = GSK618334dose 4, G = GSK618334 dose 6, I= GSK618334 dose 8. In each dosing period 2 subjects will receive placebo and 8 subjects will receive GSK618334. Subjects within a cohort will have a washout period of at least two weeks from last dose before receiving another dose.
  Interventions: Drug: GSK618334; Drug: GSK618334 matching placebo tablets

INTERVENTIONS:
Drug: GSK618334 — GSK618334 will be available as white to off-white coated tablets. GSK618334 will be swallowed with 250 milliliters (mL) of water.
Drug: GSK618334 matching placebo tablets — GSK618334 placebo tablets visually match the active GSK618334 tablets and contain the same excipients except for the omission of the active ingredient. GSK618334 matching placebo will be swallowed with 250 mL of water.

SUMMARY:
GSK618334 is being developed as an innovative treatment for substance dependence and potentially other compulsive behavioral disorders. This study will evaluate the safety, tolerability and pharmacokinetics of single doses of GSK618334 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subject, aged between 18 and 50 years of age inclusive.
* Body weight ≥50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive.
* Healthy as judged by a responsible physician. No clinically significant abnormality identified on the medical, psychiatric or laboratory evaluation, including 12-lead ECG and 24 hour Holter ECG. A subject with a clinical abnormality or laboratory parameter(s) outside the reference range for this age group may be included only if the Investigator considers the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Signed and dated written informed consent prior to participation in the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* The subject has a positive pre-study urine drug screen including alcohol at the screening visit and/or prior to receiving the first dose of study medication. Drugs that will be screened for are amphetamines, barbiturates, cocaine, opiates, cannabinoids, methadone, benzodiazepines, phencyclidine (PCP) and cotinine. If any of these tests are positive the investigator may re-test the subject and the subject may be included if the re-test is negative.
* A positive pre-study Hepatitis B surface antigen, Hepatitis C antibody, or HIV 1/2 result at the screening visit.
* Abuse of alcohol defined as an average weekly intake of greater than 28 units or an average daily intake of greater than 4 units.
* The subject has clinically significant elevations in liver function tests (LFT) that are elevated above the reference range at pre-study screening and remain elevated with a repeat LFT, and/or prior to receiving the first dose of study medication.
* Consumption of grapefruit juice or grapefruit within 7 days prior to receiving the first dose of study medication.
* Any subject who is not prepared to eat the standard meals provided by the Clinical Pharmacology Research Unit (CPRU) during the study.
* Participation in a clinical trial with a new chemical entity within 4 months before the first dose of study medication or marketed compound within 3 months before receiving the first dose of study medication.
* Use of prescription or non-prescription drugs, including, over the counter remedies, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to receiving the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Loss of more than 600mL blood during the 120 days before study start.
* History or presence of allergy to the study drug or drugs of this class, or a history of other allergy that, in the opinion of the physician responsible, contraindicates his participation in the study.
* History of regular use of tobacco- or nicotine-containing products within 6 months of the start of the study (i.e., from Screening Visit 1).
* An unwillingness of the male subject to use condoms or practise abstinence to prevent exposure of a female partner to semen from the start of the study (i.e., from Screening Visit 1) until 90 days after the study treatment has ended.
* History of psychiatric disorder either Axis I or II by DSM-IV.
* History or presence of respiratory illnesses, gastrointestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* The subject has a screening ECG with values outside of ranges defined in the protocol.
* The subject has a screening heart rate <50 or >100 bpm and a systolic blood pressure >140 and <100 mmHg and a diastolic blood pressure >90 and <60 mmHg in the semi-supine position.
* The subject has a reduction in systolic blood pressure of 20 mmHg or more, or a reduction in diastolic blood pressure of 10 mmHg or more on standing compared to the supine measurement at screening.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject is unable to abstain from strenuous physical activity for 24 h prior to the screening visit and for 24 h prior to admission for each treatment period.
* Inability of the subject to be successfully trained in tests of cognition prior to receiving the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06-28 (Actual); Primary Completion 2007-10-04 (Actual); Study Completion 2007-10-04 (Actual)

PRIMARY OUTCOMES:
Safety measures: ECG, Vital Signs, Adverse Events | for 48 hours after dosing.
PK measures: Blood sampling for GSK598809 | for up to 96hr post dose

SECONDARY OUTCOMES:
Tests on cognition (thinking) | for 48 hours after dosing
Movement rating scales | pre-dose, 2, 4 and 24 hours post-dose on Day 1
Prolactin, TSH and GH | pre-dose, 1, 2, 4, 8 and 24 hours post-dose on Day 1
Psychological assessments | pre-dose, up to 48 hours post-dose
Cognitive/Impulsivity tests | pre-dose, 2, 7 and 24 hours post-dose on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

REFERENCES:
- See also: Results for study DBU107640 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/DBU107640?search=study&search_terms=DBU107640#rs